CLINICAL TRIAL: NCT01416909
Title: Managing Medication-induced Constipation in Cancer: A Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MCC-15712
Record Dates: First submitted 2011-08-11; First posted 2011-08-15 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2015-03

CONDITIONS: Constipation
Keywords: Medication-induced; Constipation in Cancer
MeSH Terms: conditions — Constipation | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dose Intervention - Opioid (Active Comparator): Laxative Treatment: Participants Receiving Opioids for the Treatment of Pain. Participants will be taken off any laxative preparation they may already be on and will be put on laxative treatment based on the Constipation Treatment Protocol. The dose of laxative will be based on the dose of the opioid pain medication they are receiving.
  Interventions: Other: Laxative Treatment; Other: Assessment Questionnaires
- Assessment Intervention - Opioid (Active Comparator): Laxative Treatment: Participants Receiving Opioids for the Treatment of Pain. Participants will be taken off any laxative preparation they may already be on and will be put on laxative treatment based on the Constipation Treatment Protocol. The dose of laxative will be determined based on their severity of constipation.
  Interventions: Other: Laxative Treatment; Other: Assessment Questionnaires
- Control Group - Opioid (Other): Standard of Care: Participants Receiving Opioids for the Treatment of Pain will receive their usual care at Moffitt while participating in weekly assessments. After participation in the study is complete, participants will be offered the same protocol that is given to patients in the treatment groups.
  Interventions: Other: Standard of Care; Other: Assessment Questionnaires
- Assessment Intervention - Vinca Alkaloid (Active Comparator): Laxative Treatment: Participants Receiving a Specific Type of Chemotherapy (vinca alkaloids). Vinca alkaloids include medication such as Vincristine, Vinblastine, or Vinorelbine. Participants will be taken off any laxative preparation they may already be on and will be put on laxative treatment based on the Constipation Treatment Protocol. The dose of laxative will be based on their level of constipation.
  Interventions: Other: Laxative Treatment; Other: Assessment Questionnaires
- Control Group - Vinca Alkaloid (Other): Standard of Care: Participants Receiving a Specific Type of Chemotherapy (vinca alkaloids). Vinca alkaloids include medication such as Vincristine, Vinblastine, or Vinorelbine. Patients will receive standard of care while participating in weekly assessments. After participation in the study is complete, participants will be offered the same protocol that is given to patients in the treatment groups.
  Interventions: Other: Standard of Care; Other: Assessment Questionnaires

INTERVENTIONS:
Other: Laxative Treatment — Participants will be taken off any laxative preparation they may already be on. Patients will be put on laxative treatment based on the Constipation Treatment Protocol.
  Other Names: constipation treatment
  Arms: Assessment Intervention - Opioid; Assessment Intervention - Vinca Alkaloid; Dose Intervention - Opioid
Other: Standard of Care — Participants will receive their usual care at Moffitt while participating in weekly assessments. After participation in the study is complete, participants will be offered the same protocol that is given to patients in the treatment groups.
  Arms: Control Group - Opioid; Control Group - Vinca Alkaloid
Other: Assessment Questionnaires — Constipation Assessment Scale (CAS), Laxative Interview (based on Laxative Diary completed by patients), Memorial Symptom Assessment Scale (MSAS), Functional Assessment of Cancer Therapy-General (FACT-G).

SUMMARY:
The purpose of this research is to evaluate the effectiveness of the Constipation Treatment Protocol and to test whether management according to dose of constipation-inducing medications or according to on-going assessment is most effective.

DETAILED DESCRIPTION:
Patients will undergo a baseline assessment during their regular outpatient visit. With their permission, the investigators will audio record this visit for quality control. After the study, the recordings will be erased. Patients will be asked to complete 4 questionnaires. The investigators will collect contact information so that the follow-up assessments can be done by phone.

ELIGIBILITY:
Inclusion Criteria:

* The study sample will consist of patients who are receiving outpatient care at the Moffitt Cancer Center.
* Patients will be identified as those who have a diagnosis of cancer and are being treated with either opioids or vinca alkaloids,
* are adults (or children 18-21 years old),
* either male or female,
* able to read and understand English,
* and able to pass screening with the Short Portable Mental Status Questionnaire and Karnofsky Performance Status Scale.

Exclusion Criteria:

* Patients will be excluded: if they have non-melanoma skin cancer or colorectal or gynecological cancer as their primary diagnosis;
* if they are excessively debilitated or deemed unlikely to survive for the eight weeks of the data collection period;
* if they are unable to read and understand English;
* if they have an ostomy that changes bowel function;
* if they have a current peritoneal catheter;
* if they have had abdominal surgery within the past six weeks;
* or have a disease process suggestive of mechanical obstruction (tumor or adhesion);
* if they have a history of chronic bowel disease (including irritable bowel syndrome, chronic constipation prior to cancer onset, Crohn's disease, ulcerative colitis or diarrhea as a result of radiation to the pelvis), or report chronic laxative use prior to cancer onset.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2008-11; Primary Completion 2013-08 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Phase I - Record Constipation Incidence and Symptoms | 18 months
  To identify the incidence, severity, distress and trajectory of constipation in cancer patients receiving opioids over an eight week period and to evaluate the relationships between constipation intensity and opioid dose.
  To identify the incidence, severity, distress and trajectory of constipation in groups of cancer patients who may be at risk due to vinca alkaloids (vincristine. vinblastine. vinorelbine and vindesine) over an eight week period and to evaluate the relationship between constipation intensity and vinca alkaloid dose.

SECONDARY OUTCOMES:
Phase II - Number of Participants With Desired Effect - Patients with Medication-induced Constipation | 2 years, 3 months
  To test the efficacy of a Constipation Treatment Protocol in patients with medication-induced constipation.
Phase II - Best Determination of Laxative Dose - Patients with Medication-induced Constipation | 2 years, 3 months
  To test whether laxative dose is best determined based on on-going assessment or on opioid dose.
  To test whether laxative dose is best determined based on on-going assessment or on vinca alkaloid dose.

CONTACTS AND LOCATIONS:
Overall Officials: Susan McMillan, Ph.D., RN, Principal Investigator — University of South Florida
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States